CLINICAL TRIAL: NCT04232020
Title: A Retrospective Validation of Idylla Microsatellite Instability Testing Versus Mismatch Repair Immunohistochemistry in Gastric Adenocarcinoma Biopsies
Brief Title: A Retrospective Validations Microsatellite Instability (MSI) Testing v Mismatch Repair (MMR) in Gastric Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2019.RCHT.107
Record Dates: First submitted 2020-01-06; First posted 2020-01-18 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — DNA Mismatch Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — formalin fixed paraffin processed tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mismatch repair — MSI testing using Biocartis Idylla and MMR immunohistochemistry

SUMMARY:
To compare the Idylla microsatellite instability test versus mismatch repair immunohistochemistry (IHC) in gastric adenocarcinoma.

DETAILED DESCRIPTION:
Gastric adenocarcinoma is a common form of cancer which is associated with a poor prognosis. Up to 22% of gastric adenocarcinomas arise via the microsatellite instability (MSI) / mismatch repair (MMR) pathway. These cases can be detected either by mismatch repair immunohistochemistry (IHC) or microsatellite instability testing. Detection of mismatch repair deficiency or microsatellite instability is important because patients with this type of gastric adenocarcinoma are shown to benefit from a different therapeutic approach. High concordance between mismatch repair immunohistochemistry and microsatellite instability testing has already been demonstrated. The implementation of either method is largely based on local availability. The Idylla MSI test presents a novel method of establishing MSI status in comparison to pre-existing MSI testing platforms. The Idylla MSI tests uses a fully automated, ultra-rapid system that can work on formalin-fixed, paraffin embedded tissue with no need for preceding DNA extraction. Implementation of the Idylla MSI test could reduce reporting turnaround times and requires less technical expertise to perform in comparison to other platforms.

The investigators department does not currently have the facilities to perform MSI testing on any platform, so the advantages of introducing the Idylla MSI test would also include the generic advantages of MSI testing. These advantages include: the ability to quickly check cases shown to have possible MMR loss on IHC (i.e. equivocal cases) with MSI testing; and providing an alternative to MMR IHC for screening of Lynch syndrome, reducing the burden on reporting pathologists and reduce the inter-observer variability associated with IHC interpretation.

The Idylla MSI test already demonstrates high concordance with other MSI testing platforms but has yet to be compared to the department's accepted standard of MMR IHC. This project aims to compare the Idylla MSI test to in-house MMR IHC to establish whether the two methods are concordant in reporting MMR / MSI status in gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient consent
* Adequate tissue including adequate tumour burden
* Diagnosis of adenocarcinoma in this biopsy

Exclusion Criteria:

* No patient consent
* Inadequate tissue or block not present in archive
* No adenocarcinoma in biopsy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study involves the use of pre-existing tissue samples and has no patient participation apart from the use of the existing sample.
  Only samples that have been identified with an adenocarcinoma diagnosis and with an adequate amount of tissue sample available will be used in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Idylla MSI test using Idylla MSI Cartridges to assess suitability | 6 months
  MMR IHC panels will be passed to the histopathology team for interpretation. Cases will be interpreted and results will be determined by either a) loss of staining or b) no loss of staining of any individual antibody

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jones, Principal Investigator — Senior Biomedical Scientist
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided